CLINICAL TRIAL: NCT05949671
Title: Evaluation of the Effect of Gluten-Free Diet and Mediterranean Diet on the Autoimmune System in Patients With Hashimoto's Thyroid
Brief Title: Evaluation of the Effect of Gluten-Free Diet and Mediterranean Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACU-BES-SBF-MUTLUTUCEULKER-001
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Hashimoto Thyroiditis; Hashimoto Disease
Keywords: Mediterranean diet; Mediterranean gluten-free diet; Gluten-free diet; hashimoto
MeSH Terms: conditions — Hashimoto Disease | interventions — Diet, Gluten-Free

STUDY DESIGN:
Intervention Model Description: doctoral thesis including case and control groups
Who Masked: Participant
Masking Description: patients do not know which group they belong to and other groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mediterranean groups (Experimental): This study is a prospective, single-blind study including case and control groups. Before the study started, participants were informed about the benefits and risks of the study. Participants were randomly divided into four different groups (MD, GFD, MGFD and control group). The intervention groups (MD group (n=10)) were administered weekly diets by a dietitian for 12 weeks according to individual-specific and daily energy needs and weight loss was not targeted. Patients were interviewed weekly to assess adherence to the study protocol and food consumption was recorded at each interview; those who complied with the weekly planned menus by less than eighty percent were excluded from the study.
  Interventions: Other: mediterranean, gluten-free and mediterranean gluten-free diet intervention
- Gluten-Free groups (Experimental): This study is a prospective, single-blind study including case and control groups. Before the study started, participants were informed about the benefits and risks of the study. Participants were randomly divided into four different groups (MD, GFD, MGFD and control group). The intervention groups (GFD (n=10)) were administered weekly diets by a dietitian for 12 weeks according to individual-specific and daily energy needs and weight loss was not targeted. Patients were interviewed weekly to assess adherence to the study protocol and food consumption was recorded at each interview; those who complied with the weekly planned menus by less than eighty percent were excluded from the study.
  Interventions: Other: mediterranean, gluten-free and mediterranean gluten-free diet intervention
- Mediterranean Gluten-Free groups (Experimental): This study is a prospective, single-blind study including case and control groups. Before the study started, participants were informed about the benefits and risks of the study. Participants were randomly divided into four different groups (MD, GFD, MGFD and control group). The intervention groups (MGFD (n=10)) were administered weekly diets by a dietitian for 12 weeks according to individual-specific and daily energy needs and weight loss was not targeted. Patients were interviewed weekly to assess adherence to the study protocol and food consumption was recorded at each interview; those who complied with the weekly planned menus by less than eighty percent were excluded from the study.
  Interventions: Other: mediterranean, gluten-free and mediterranean gluten-free diet intervention
- control group (No Intervention): Patients in the control group (n=10) did not receive any special dietary intervention.

INTERVENTIONS:
Other: mediterranean, gluten-free and mediterranean gluten-free diet intervention — This study is a prospective, single-blind study including case and control groups. Before the study started, participants were informed about the benefits and risks of the study. Participants were randomly divided into four different groups (MD, GFD, MGFD and control group). The intervention groups (MD group (n=10), GFD (n=10), MGFD (n=10)) were administered weekly diets by a dietitian for 12 weeks according to individual-specific and daily energy needs and weight loss was not targeted. Patients in the control group (n=10) did not receive any special dietary intervention. Patients were interviewed weekly to assess adherence to the study protocol and food consumption was recorded at each interview; those who complied with the weekly planned menus by less than eighty percent were excluded from the study.
  Arms: Gluten-Free groups; Mediterranean Gluten-Free groups; Mediterranean groups

SUMMARY:
Background: Hashimoto's Thyroiditis is an autoimmune disease that attacks thyroid cells through cell- and antibody-mediated immune processes and is characterized by the production of thyroid autoantibodies. In hashimoto, antithyroid peroxidase antibodies are increased and thyroid stimulating hormone levels are elevated. A gluten-free diet regulates thyroid autoimmunization by decreasing the concentration of antibodies. The Mediterranean diet also reduces disease-related oxidative stress parameters in patients with hashimoto's thyroid due to its anti-inflammatory effects.

Aims: To evaluate the short-term effects of Mediterranean, gluten-free and Mediterranean gluten-free dietary patterns on thyroid function and autoantibody levels of patients.

Study Design: Prospective, single-blind randomized controlled trial including case and control groups Methods: The 40 patients with hashimato thyroiditis included in the study were randomly divided into 4 different groups as gluten-free, Mediterranean, Mediterranean gluten-free and control group for 12 weeks. Thyroid function tests and autoantibody levels were analyzed at the beginning and end of the study. In addition, anthropometric measurements were taken at the beginning and end of the study and food consumption records and food consumption frequencies were evaluated.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the short-term effects of Mediterranean (MD), Gluten Free (GFD) and Mediterranean Gluten Free (MGFD) dietary patterns on the autoimmune system in patients with Hashimoto's Thyroiditis. The study was planned as a prospective single-blind study including case and control groups and 40 women with hashimoto participated. Study participants were not taking medication or supplements to better evaluate the effect of the nutritional intervention on thyroid function. Participants were divided into 4 groups as MD, GFD, MGFD nutrition intervention groups and control group. At the beginning of the study and after three months of nutritional intervention, anthropometric measurements, body composition analysis, thyroid function tests were performed, food consumption records and food consumption frequencies were taken. Weekly menus were planned and the compliance of the individuals with the nutritional intervention applied for three months was evaluated. In this study, the decrease in antibody levels and changes in thyroid function tests were evaluated as short-term effects of the nutritional intervention. Long-term studies evaluating the changes on antibodies with nutritional intervention are needed.

ELIGIBILITY:
Inclusion Criteria:

* To apply to the Internal Diseases (Internal Medicine) outpatient clinic, to be diagnosed with hashimato thyroid (HT) by a physician and to be between the ages of 18-65,
* No diagnosis of any autoimmune system disease other than HT that may adversely affect the study,
* No symptoms of celiac disease and no diagnosis,
* Not following a gluten-free diet in the last three months,
* Not being diagnosed with an eating behaviour disorder,
* Not having any communication problems,
* Signing the informed consent form,
* Having had a thyroid ultrasound within the last six months,
* Elevated anti -TPO (>5.61 IU/ml) and anti Tg (>4.11 IU/ml),
* To have TSH, Free T3 and Free T4 tests performed,
* Body Mass Index to be in the range of 18.5 kg/m2 - 30 kg/m2 <,
* Not losing 5% and/or more body weight in the last month

Exclusion Criteria:

* - Under 18 years of age and over 65 years of age,
* Having thyroid disease other than HT,
* Having a diagnosis of autoimmune system disease other than HT that may adversely affect the study,
* Symptoms and/or diagnosis of celiac disease,
* To have been diagnosed with non-celiac gluten sensitivity,
* Following a gluten-free diet within the last three months,
* A diet therapy that has an effect on the autoimmune system within the last three months,
* Being diagnosed with eating behaviour disorder,
* Having any communication problems,
* Not signing the informed consent form,
* Failure to adapt to the work during the working period, to be in a situation/behaviour that may adversely affect the work,
* To have applied any nutritional intervention during the last three months prior to the study,
* Being pregnant or breastfeeding,
* Taking supplements such as selenium, zinc, vitamin D and/or iodine, which may affect the course of the study,
* To have received cancer treatment and / or to be receiving cancer treatment,
* Having other endocrine or metabolic diseases (e.g. diabetes, cardiovascular diseases),
* Diagnosed with a disease lasting more than 4 months in the last 12 months and other specialised dietary / compositionally different dietary patterns (e.g. high protein, ketogenic, low energy content < 1000 kcal/day),
* Body Mass Index <18.5 kg/m2 or BMI≥30 kg/m2,
* Loss of 5% and/or more body weight in the last month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with hashimoto's thyroiditis
Enrollment: 40 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Effect of Gluten-Free Diet and Mediterranean Diet on the Autoimmune System in Patients with Hashimoto's Thyroid | May 2021-June2022
  Diet group (MD group (n=10)) was administered weekly diets for 12 weeks by a dietitian according to personalised and daily energy needs and weight loss was not targeted.

OTHER OUTCOMES:
Evaluation of the Effect of Gluten-Free Diet and Mediterranean Diet on the Autoimmune System in Patients with Hashimoto's Thyroid | May 2021-May 2022
  Diet group (MD group (n=10)) was administered weekly diets for 12 weeks by a dietitian according to personalised and daily energy needs and weight loss was not targeted.

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Tuçe Ülker, Dr, Principal Investigator — Acibadem University
Locations (1):
- Istınye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided